CLINICAL TRIAL: NCT04512391
Title: Analgesic Efficacy of Erector Spinae Plane Block After Breast Cancer Surgery
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, ersin sönmez, Research Assistant, TC Erciyes University
Other Study IDs: 2020/134
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Postoperative Pain; Breast Cancer
Keywords: Erector spinae plane block; breast cancer; surgery; postoperative pain; analgesic
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Erector Spinae: patients who are administered ultrasound guided ESPB at T4 vertebrae level with long acting local anesthetic (%0,25 bupivacaine) and followed up with patient controlled analgesia device and all records about aforementioned data is completely available.
  Interventions: Procedure: Ultrasound guided Erector Spinae Plane Block (ESPB)
- Control: patients who are not administered any regional analgesic technique and followed up with patient controlled analgesia device and all records about aforementioned data is completely available.

INTERVENTIONS:
Procedure: Ultrasound guided Erector Spinae Plane Block (ESPB) — Ultrasound guided ESPB is applied at T4 vertebrae level, 3 cm lateral to mid-line where transverse process lies. After identification of transverse process, needle is advanced in plane and real time visualisation on ultrasound screen. When bonny contact is encountered, normal saline is injected for verification of placement, then, 25 ml %0,25 bupivacaine is injected plane between transverse process and erector spinae muscles.
  Groups: Erector Spinae

SUMMARY:
Erector spinae plane block(ESPB), which is firstly used for thoracic neuropathic pain, is newly developed and highly promising fascial plane block for providing postoperative analgesia for a great deal of surgeries including breast surgery. The investigators aim to study efficacy of ESPB for patients who undergone breast cancer surgery and is expected to benefit from opioid-sparing effect of this technique.

DETAILED DESCRIPTION:
This is a retrospective, single-center clinical trial to evaluate analgesic efficacy of Erector spinae plane block (ESPB) after breast cancer surgery. Participant's demographics and medical history, type and extent of surgery, systemic opioid and non-opioid analgesic consumptions, hemodynamic variables and adverse events during and first 24 hours after surgery. After operation, pain scores at first 24 hours, 1., 3., and 6. month will be obtanied from surgical ward and pain clinic registires. patient controlled analgesia device usage history will be obtained from device database at our clinic.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients undergoing breast surgery for breast cancer
* Becoming available of complete records about study data

Exclusion Criteria:

* ASA III-IV patients
* missing records about study data

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: all patients undergoing breast surgery for breast cancer between September 2018 and December 2019 were included in our study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | First 24 hours after surgery
  all patients were given 0.05 mg/kg morphine iv and 1 gr paracetamol 30 minutes before end of surgery and in the recovery room, a patient- controlled analgesia device containing morphine 0.5 mg/ml, set to deliver a 1mg bolus dose of morphine with an 10 min lockout time. Total morphine consumption during the 24 hours postoperative period will recorded at 5 times intervals ( 2, 4, 6, 12, 24 hours).
Verbal Analog Pain Scores on rest and movement | First 24 hours after surgery, at 1., 3., 6. month
  A Research assistant, blinded to the group allocation, interviewed patients and collected data at 5 times intervals ( 2, 4, 6, 12, 24, hours) in the 24 hours postoperatively. Patients were asked to rate their pain using verbal analog scale, where 0= no pain and 10= worst pain possible.

SECONDARY OUTCOMES:
Demographic Data | First 24 hours after surgery
  Age, sex, medical history, BMI, ASA (American Society of Anesthesiologists) status, Duration and type of surgery were recorded
Blood Pressures | during and first 24 hours after surgery
  systolic, diastolic and mean arterial blood pressures as mmHg
Heart Rate | during and first 24 hours after surgery
  Heart rate as beat per minute (BPM)
incidence of adverse effects (like nausea and vomiting) | First 24 hours after surgery
  incidence of nausea and vomiting during the 24 hours postoperative period was recorded recorded at 5 times intervals ( 2, 4, 6, 12, 24 hours)
Rescue analgesic requirement | First 24 hours after surgery
  number of request and dosages of non opioid analgesics used for VAS equal or greater than 5 or patient request.

CONTACTS AND LOCATIONS:
Overall Officials: ersin SÖNMEZ, Principal Investigator — Research Asisstant
Locations (1):
- TC erciyes university, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005